CLINICAL TRIAL: NCT00768794
Title: A Trial Using Acidophilus for the Treatment and Prevention of Oral Candidiasis in Head and Neck Cancer Patients Undergoing Radiation Therapy
Brief Title: Acidophilus for the Treatment and Prevention of Oral Candidiasis in Patients Undergoing Radiation Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Summa Health System (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Acidophilus
Record Dates: First submitted 2008-10-07; First posted 2008-10-08 (Estimated); Last update posted 2013-05-31 (Estimated); Status verified 2013-05

CONDITIONS: Oral Candidiasis
Keywords: thrush
MeSH Terms: conditions — Candidiasis, Oral | interventions — Lacteol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Acidolphilus (Active Comparator): In the first part of the study, two participants will begin radiation therapy. When signs and symptoms of thrush are noted, such as smooth, creamy, white/yellow coating and/or patches on the tongue and inside of their mouth that are painful, subjects will begin taking acidophilus capsules twice each day until the last day of radiation therapy.
  Interventions: Dietary Supplement: Acidophilus; Dietary Supplement: Acidolphilus

INTERVENTIONS:
Dietary Supplement: Acidophilus — Use of Acidophilus in the first part of the study, two participants will begin radiation therapy. When signs and symptoms of thrush are noted, such as smooth, creamy, white/yellow coating and/or patches on the tongue and inside of their mouth that are painful, subjects will begin taking acidophilus capsules twice each day until the last day of radiation therapy.
  The second part of the study is to determine if acidophilus is effective in preventing oral candidiasis (thrush) during radiation therapy to the head and neck region.
Dietary Supplement: Acidolphilus — The second part of the study is to determine if acidophilus is effective in preventing oral candidiasis (thrush) during radiation therapy to the head and neck region.

SUMMARY:
The purpose of this study is to determine the effectiveness of using acidophilus to treat oral candidiasis (thrush) caused by radiation therapy to the head and neck region.

This study will conducted in two parts. In the first part of the study, two participants will begin radiation therapy. When signs and symptoms of thrush are noted, such as smooth, creamy, white/yellow coating and/or patches on the tongue and inside of your mouth that are painful, you will begin taking acidophilus capsules twice each day until the last day of radiation therapy.

The second part of the study is to determine if acidophilus is effective in preventing oral candidiasis (thrush) during radiation therapy to the head and neck region. In the second part of the study three participants will take acidophilus capsules twice each day beginning on the first day of radiation therapy and continuing until the last day of radiation therapy.

DETAILED DESCRIPTION:
To determine if Lactobacillus acidophilus ,Ritzman Natural Health Acidophilus supplements given twice daily during radiation treatments to the head and neck region after the development of oral thrush is an effective treatment for oral candidiasis.

To determine if Lactobacillus acidophilus ,Ritzman Natural Health Acidophilus supplements given twice daily beginning on the first day of radiation treatments to the head and neck region prevents the development of oral thrush.

To assess subjective and objective response of oral candidiasis treated with Lactobacillus acidophilus ,Ritzman Natural Health Acidophilus supplements.

To assess the efficacy of Lactobacillus acidophilus ,Ritzman Natural Health Acidophilus supplements in preventing oral candidiasis in patients receiving radiation therapy to the head and neck region.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically (histologically or cytologically) proven diagnosis of squamous cell carcinoma of the head and neck region receiving > 50 Gy to head and neck tumor with or without concomitant chemotherapy and/or cetuximab.
* Age ≥ 18
* Karnofsky Performance Score of > 70
* History and physical examination within 8 weeks prior to registration
* Patient must sign study specific informed consent prior to study entry.

Exclusion Criteria:

* Prior invasive malignancy (except non-melanomatous skin cancer) unless disease free for a minimum of 3 years.
* Patients with carcinoma in-situ of the breast, oral cavity, or cervix are eligible.
* Prior radiotherapy to the region of the study cancer that would result in overlap of radiation therapy fields.
* Acute bacterial or fungal infection requiring intravenous or oral antibiotics at study entry
* Sjoren's syndrome
* Hypoadrenalism
* Acquired Immune Deficiency Syndrome (AIDS) based upon current CDC definition; note, however, that HIV testing is not required for entry into this protocol.
* Pregnancy or women of childbearing potential and men who are sexually active and not willing/able to use medically acceptable forms of contraception.
* Prior allergic reaction to Lactobacillus acidophilus.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2006-07; Primary Completion 2010-03 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
To determine if Lactobacillus acidophilus ,Ritzman Natural Health Acidophilus supplements given twice daily during radiation treatments to the head and neck region after the development of oral thrush is an effective treatment for oral candidiasis. | during duration of treatment of 4 weeks.

SECONDARY OUTCOMES:
To the response of oral candidiasis treated with Lactobacillus acidophilus ,Ritzman Natural Health Acidophilus supplements and to determine efficacy. | during duration of treatment of 4 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Heather Tharpe, Rn, BSN, OCN, Principal Investigator — Summa Health System; Joyce Neading, RHIT, CTR, Study Director — Summa Health System
Locations (1):
- Summa Health System, Akron, Ohio, United States